CLINICAL TRIAL: NCT05419518
Title: Palliative Dose Escalated Radiation for Painful Non-Spine Bone Metastases and Painful Non-Bone Metastases
Brief Title: Palliative Dose Escalated Radiation for Painful Non-Spine Bone Metastases and Painful Non-Bone Metas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Matthew Pierre Deek, Assistant Professor, Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152201; Pro2022000822 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Neoplasm Metastases; Metastases, Neoplasm
Keywords: Metastase; Bone Neoplasms; Dose Fractionation, Radiation
MeSH Terms: conditions — Neoplasm Metastasis; Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an, open label, single-institution, Phase II trial of palliative radiation dose escalation study for painful non-spine bone Metastases and painful non-bone metastases.
  Dose escalation with 2D/ 3D-CRT in ten fractions in non-spine bone metastases will be evaluated. The total dose will range from 40-50 Gy depending on normal tissue constraints. This dose in ten fractions will lead to BED10 of 56 - 75 Gy which is higher than the BED10 39 Gy with 30 Gy in ten fractions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palliative radiation dose escalation (Experimental): The prescribed dose is 50 Gy in 10 fractions. The total dose can be reduced to 40 Gy and the total number of fractions can be reduced to 8 fractions in non-spine metastases to achieve the normal tissue constraints.
  Interventions: Biological: EXTERNAL BEAM RADIATION
- Therapeutic benefit (No Intervention): Radiation will be delivered as per protocol. For participants experiencing unacceptable toxicity related to study treatment, yet obtaining therapeutic benefit, participants will be allowed to continue treatment, if well tolerated at the discretion of the investigator.

INTERVENTIONS:
Biological: EXTERNAL BEAM RADIATION — A minimum of three daily radiation therapy treatments are required in any given week. Any missed radiation treatments will be made up at the end of the treatment schedule, such that the total number of delivered 5 Gy fractions remains ten.
  Arms: Palliative radiation dose escalation

SUMMARY:
The investigators hypothesize that with dose escalation to 40-50 Gy in ten fractions, the complete pain response rate at one month can be increased to 40-50% in painful non-spinal bone metastases. Additionally, the investigators hypothesize that utilizing a fractionation scheme with an escalated biologically equivalent dose (BED) will result in a higher proportion of participants responding to treatment, and will also lead to more durable responses. Furthermore, the investigators hypothesize that with dose escalation to 40-50 Gy in ten fractions, the complete pain response rate at one month can be increased to 35-45% in painful non-bone metastases

DETAILED DESCRIPTION:
The purpose of this study is to prospectively evaluate dose escalation and pain response in patients with painful non-spinal bone metastases and painful non-bone metastases treated with radiation therapy.

Primary Objective:

To evaluate improvement of complete pain response rate in painful non-spine bone metastases and painful non-bone metastases with dose escalated radiation using a ten fraction radiation regimen

Secondary Objectives:

To evaluate best pain response To evaluate mean pain scores To evaluate the duration of pain response To evaluate the changes in quality-of-life following radiation To evaluate the rates of retreatment with radiation secondary to disease or symptom progression To evaluate treatment related toxicity

ELIGIBILITY:
Inclusion Criteria:

* Have provided signed informed consent for the trial
* Aged ≥18 years at the time of informed consent
* Histologic proof of malignancy
* Radiologic or histologic evidence of bone metastases or non-bone metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≥3
* Pain Score ≥ 3
* Life expectancy of six months or more
* Willing and able to comply with all aspects of the protocol
* A female participant is eligible to participate if she is not pregnant and not breastfeeding
* Woman of childbearing potential who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

* Metastasis from a highly radiosensitive tumor (eg, lymphoma, myeloma, germ cell tumor)
* Spinal metastasis
* Active compression of spinal cord/cauda equina
* Previous RT or SBRT to the same site
* > 3 sites requiring radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of participants experiencing adverse events | One month
  Number of participants experiencing adverse effects grade three or higher, as defined by Common Terminology Criteria for Adverse Effects version 5.0 (CTCAE v5.0)

SECONDARY OUTCOMES:
Severity as assessed by number of participants experiencing toxicity and adverse events | One month
  This study will utilize the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 5.0 for toxicity and Adverse Event reporting

OTHER OUTCOMES:
Pain as assessed by number of participants experiencing pain response | One month
  will be measured according to the international consensus guidelines on palliative RT13.
  Pain assessment will be based on scores in Numerical Rating Pain Scale (NRPS), Visual analog scale (VAS) and Opioid analgesic use (an oral morphine equivalent dose (OMED)) in mg.
  Complete response is defined as a pain score of 0 on a scale from 0 to 10 and without an increase in OMED medication use.
  Partial response is defined as a decline of ≥2 points in pain score without analgesic increase or a decline in use of OMED of at least 25% or more from baseline without an increase in pain.
  Pain progression (PP) is an increase of ≥2 points without a change in OMED use or an increase of 25% or more in OMED compared with baseline with the pain score stable or one point above baseline.
Quality-of-life (QOL) as assessed by the Brief Pain Inventory (BPI). Using the 16 item scale | One month
  Quality-of-life (QOL) instruments specific to participants with bone metastases or to those receiving palliative care have been developed in recent years. The Brief Pain Inventory (BPI) have shown excellent reliability and validity in assessing participants with bone metastases fourteen. BPI will be used for QOL assessment at baseline and one month after treatment.The BPI scale defines pain as follows:
  Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Deek, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (7):
- United States (7):
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - RWJBarnabas Health - Saint Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No